CLINICAL TRIAL: NCT04820660
Title: Effects of Task-oriented Progressive Resistance Strength Training and Balance Exercises in Functional Performance on Lower Limb in Individuals With Stroke
Brief Title: Task-oriented Progressive Resistance Strength Training and Balance Exercises on Lower Limb in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/19/2033 Hira Javed
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Balance; progressive resistance strength training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task oriented Strength training group (Experimental): Standing and reaching in different directions Sit-to-stand Stepping forward and backward Stepping sideways onto blocks
  Interventions: Other: Task orientated strengthening training
- Balance Training (Experimental): Stepping forward, backward, and sideways on the exercise step; Stepping over blocks of various heights; Standing up from a chair, From a sitting position on a 65-cm Swiss ball, Arms; bending the trunk forward and side to side); Performing double-legged stance Performing tandem stance Rising from a chair without the use of the arms; Walking forward and backward with a tandem walking pattern Performing single- legged stance
  Interventions: Other: Balance training exercises

INTERVENTIONS:
Other: Task orientated strengthening training — 1. Standing and reaching in different directions for objects located beyond arm's length to promote loading of the lower limbs and activation of lower limb muscles;
  2. Sit-to-stand from various chair heights to strengthen the lower limb extensor muscles;
  3. Stepping forward and backward onto blocks of various heights to strengthen the lower limb muscles;
  4. Stepping sideways onto blocks of various heights to strengthen the lower limb muscles;
  5. forward step-up onto blocks of various heights to strengthen the lower limb muscles;
  6. heel(s) raise and lower while maintaining in a standing posture to strengthen the plantar- flexor muscles.
  Each workstation was 5 min in duration for each exercise class. Each subject participated in a one-to-one therapy.
  Arms: Task oriented Strength training group
Other: Balance training exercises — 1. Stepping forward, backward, and sideways on the exercise step;
  2. Stepping over blocks of various heights;
  3. Standing up from a chair, walking four steps forward, performing a bilateral stool touch and walking backwards to the chair;
  4. Standing up from a chair, walking four steps forward, turning to the right, stepping over the exercise step, turning to the right again and walking forwards to the chair (repeat the exercise circuit in opposite direction);
  5. From a sitting position on a 65-cm Swiss ball, performing a range of motion and balance exercises (forward and backward rolling of the
  6. Arms; bending the trunk forward and side to side);
  7. Performing double-legged stance for 10 s;
  8. Performing tandem stance for 10 s;
  9. Rising from a chair without the use of the arms;
  10. Walking forward and backward with a tandem walking pattern (toes of one foot touching the heel of the foot in front);
  11. Performing single- legged stance for 10 s.
  Arms: Balance Training

SUMMARY:
Stroke is ranked as the number fifth cause of death and a main cause of disability in the United States. It affects the arteries which supply blood to and within the brain. If the blood supply to the brain is disrupted, it will not be able to receive oxygen and the nutrients which are transported by those arteries. This leads to the death of brain cells having a magnificent effect on the function of that part.

DETAILED DESCRIPTION:
This study was quasi-experimental trial, to compare the effectiveness of Progressive Resistive Strength Exercises and Balance Exercises in subjects with Stroke. Subjects with Stroke meeting the predetermined inclusion & exclusion criteria were divided into two groups using lottery method. Pre assessment was done using Berg Balance Scale, Fugl Meyer Assessment - Lower Extremity and Step Test.

Subjects in one group were treated with Progressive Resistive Strength Training and other group was treated with Balance training. Each subject received 12 treatment sessions, with 03 treatment sessions per week. Results were recorded at the end of 3rd, 6th, 9th and 12th treatment sessions. Recorded values were analysed using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic from a single stroke occurring at least a year earlier, not presently receiving any rehabilitation services,
* Participants should not be receiving any rehabilitation services
* Participants should be able to walk 10 m independently without an assistive device
* Participants should be medically stable enough to allow participation, and able to understand instructions and follow commands.

Exclusion Criteria:

* Participants with any medical condition that would prevent participation in the training program
* Participants with any uncontrolled health condition for which exercise is contraindicated.
* Participants with any tumor or neurological signs.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 4months
  Zero indicates the lowest level of function and 4 the highest level of function. The total score ranges from 0 to 56.
Fugl Meyer Assessment Lower Extremity | 4 months
  Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Background] van der Worp HB, van Gijn J. Clinical practice. Acute ischemic stroke. N Engl J Med. 2007 Aug 9;357(6):572-9. doi: 10.1056/NEJMcp072057. No abstract available. PMID 17687132
- [Background] Andersen KK, Olsen TS, Dehlendorff C, Kammersgaard LP. Hemorrhagic and ischemic strokes compared: stroke severity, mortality, and risk factors. Stroke. 2009 Jun;40(6):2068-72. doi: 10.1161/STROKEAHA.108.540112. Epub 2009 Apr 9. PMID 19359645
- [Background] Albers GW, Caplan LR, Easton JD, Fayad PB, Mohr JP, Saver JL, Sherman DG; TIA Working Group. Transient ischemic attack--proposal for a new definition. N Engl J Med. 2002 Nov 21;347(21):1713-6. doi: 10.1056/NEJMsb020987. No abstract available. PMID 12444191
- [Background] Lovett JK, Dennis MS, Sandercock PA, Bamford J, Warlow CP, Rothwell PM. Very early risk of stroke after a first transient ischemic attack. Stroke. 2003 Aug;34(8):e138-40. doi: 10.1161/01.STR.0000080935.01264.91. Epub 2003 Jul 10. PMID 12855835